CLINICAL TRIAL: NCT05325918
Title: HIF-1 Alpha, VEGF and MMP-8 Levels in Peri-implant Crevicular Fluid of Smokers Versus Non Smokers
Brief Title: HIF-1 Alpha, VEGF and MMP-8 Levels in PICF of Smokers Versus Non Smokers
Status: Completed | Type: Observational
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Sarah Elkot, Lecturer of Oral Medicine, Periodontology and Diagnosis, Faculty of Oral and Dental Medicine, Future University in Egypt, Cairo, Egypt., Future University in Egypt
Other Study IDs: FUE13
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Peri-Implantitis
Keywords: gingival crevicular fluid; Smoking; inflammation
MeSH Terms: conditions — Peri-Implantitis; Smoking; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peri-implant crevicular fluid samples collected using periopaper strips
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Smoking is a major risk factor for developing peri-implantitis so the current study is comparing inflammatory markers in smokers versus non smokers to know if they have a potential role in pathogenesis of peri-implantitis

DETAILED DESCRIPTION:
Peri -implant crevicular fluid was obtained from seven smoker patients and then compared to peri-implant crevicular fluid from seven non smoker individuals.

The peri-implant crevicular fluid was obtained using periopaper strips then analyzed using ELISA kits of these markers; HIF-1 Alpha, VEGF and MMP-8

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients
* Individuals with restored implants placed one year or more before study enrollment
* Both genders
* Age range 20-50 years old

Exclusion Criteria:

* Pregnant Females
* Lactating females

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Smoker patients with restored implants
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-08-29 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Measurement of levels of HIF-1 Alpha, VEGF and MMP-8 in peri-implant crevicular fluid | Baseline
  Markers collected using periopaper strips

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Elkot, Lecturer, Principal Investigator — Lecturer of Oral Medicine and Periodontology
Locations (1):
- Faculty of oral and dental medicine,FUE, Cairo,Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided